CLINICAL TRIAL: NCT00693212
Title: Further Studies of Attention Deficit Disorder - Residual Type
Brief Title: Further Studies of Attention Deficit Disorder - Residual Type (RT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Paul H. Wender MD Director Mood Disorders Clinic, University of Utah; Mood Disorders Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 1491
Expanded Access: Available
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Adult; crossover; randomized; Long-term; Open-label; methylphenidate; Social adjustment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Social Adjustment | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- a (Experimental): This arm was only open to subjects entering the second, open-label phase. All subjects were given open-label methylphenidate. Dosing was flexible.
  Interventions: Drug: methylphenidate
- MPH (Experimental): This is the active treatment arm of the double-blind placebo controlled phase. Patients were begun at 10 mg t.i.d. and the dose increased as necessary until a maximum dose of 60 mg/day was administered. Frequency could be increased and some patients had dosage schedules of 4 to 6 times per day
  Interventions: Drug: methylphenidate
- PBO (Placebo Comparator): This 2 week arm is the placebo part of the crossover design. Subjects receive placebo in a manner similar to the MPH arm. It lasts 2 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylphenidate — Dosing was flexible and dependent on clinical judgement, AEs and treatment response.
  Other Names: ritalin
  Arms: a
Drug: methylphenidate — Patients were begun at 10 mg t.i.d. and the dose increased as necessary until a maximum dose of 60 mg/day was administered. Frequency could be increased and some patients had dosage schedules of 4 to 6 times per day
  Other Names: ritalin
  Arms: MPH
Drug: placebo — Dosing is identical to the MPH arm except that the pills will contain no active medication.
  Arms: PBO

SUMMARY:
The first phase was a double-blind crossover design of methylphenidate in the treatment of adult ADHD. The second phase consisted of an open-label extension trial of methylphenidate in adult ADHD. It was hypothesized that methylphenidate would prove more effective than placebo in treating ADHD symptoms during the first phase. It was also hypothesized that methylphenidate responders from the double-blind trial would continue to benefit from treatment in the second phase. Improvement would include both ADHD symptoms and social adjustment.

DETAILED DESCRIPTION:
All patients received a single-blind week on placebo, followed by a double-blind random assignment crossover trial of methylphenidate and placebo, with each double-blind phase lasting two weeks. Subjects who experienced moderate or marked improvement on methylphenidate would be allowed to enter a long-term, open-label trial. ADHD symptom severity was measured monthly by a structured interview, the Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADDS), Clinical Global Impression - Improvement (CGI-I) and Global Assessment of Functioning (GAF). Social functioning was assessed by the clinician administered version of the Weissman Social Adjustment Scale (WSAS). Dosing was determined by clinical judgement, symptom improvement and AEs.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-55 years; male and female; met "Utah Criteria" for adult ADHD; 95th or higher percentile on the Parent Rating Scale and/or the Wender Utah Rating Scale;

Exclusion Criteria:

* Patients with other axis-I and axis-II diagnoses were excluded as were patients with significant medical problems.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 1986-02; Primary Completion 1994-11 (Actual); Study Completion 1994-11 (Actual)

PRIMARY OUTCOMES:
Wender-Reimherr Adult Attention Deficit Disorder Scale | Monthly

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement | monthly
The Global Assessment of Functioning (GAF). | monthly
The Weissman Social Adjustment Scale (WSAS) | At termination

CONTACTS AND LOCATIONS:
Overall Officials: Paul H Wender, MD, Principal Investigator — University of Utah
Locations (1):
- Univ of Utah, School of Medicine, Mood Disorders Clinic, Salt Lake City, Utah, United States